CLINICAL TRIAL: NCT06585280
Title: Investigating the Effect of Assistive Device Use on Patient Satisfaction
Brief Title: Assistive Device Satisfaction
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yılmaz, Research Assistant (Orthotist and Prosthetist), Istanbul Medipol University Hospital
Other Study IDs: E-10840098-202.3.02-3739
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Assistive Technology; Orthosis; Prosthesis; Device
Keywords: assistive device; orthosis; prosthesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- orthosis users
  Interventions: Other: No intervention
- prosthesis users
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Assistive devices are of critical importance for the independence and participation of disabled individuals in society and there is an increasing interest in them today. When the literature is examined, it is seen that there are few studies evaluating the use of orthotic and prosthetic assistive devices in terms of patient satisfaction. The aim of this study is to investigate the satisfaction of individuals using assistive devices in a multifaceted way.

DETAILED DESCRIPTION:
Assistive devices are medical devices designed to support the individuals functions and increase their activities. Assistive devices are of critical importance for the independence and participation of disabled individuals in society and are of increasing interest today. The use of assistive devices is a process consisting of different steps to increase the individuals participation in daily life activities.

Although assistive devices cannot completely eliminate disability, they can increase independence by reducing negative effects. There are many problems encountered in the selection of assistive devices. The problems encountered include the cost of the assistive device, the necessary application training, service delivery, environmental factors, age, gender, level of disability, and the type of device used. The success of assistive device rehabilitation is affected by many factors such as the duration and correct use of the device by the individual, their attitude towards the assistive device, their participation in treatment, and their expectations.

In low-income countries, disabled individuals have the right to access affordable, available assistive devices such as prosthetics and orthotic services according to the Convention on the Rights of Persons with Disabilities. Prosthetic and orthotic services are limited in low-income countries. In order to improve mobility and ensure greater participation of people with physical disabilities and amputees in society, assistive devices should be increased and user satisfaction should be investigated. In todays prosthetic and orthotic field, low-cost devices need to be developed and the multi-faceted satisfaction of users needs to be evaluated in terms of improvements in rehabilitation programs. Test batteries are frequently preferred in the evaluation of user satisfaction in orthosis and prosthetic rehabilitation. Generally, surveys based on individuals; expectations, satisfaction, experiences during daily life and statements of the individual regarding their assistive device are preferred. When the literature is examined, it is seen that there are few studies evaluating the use of orthosis and prosthetic assistive devices in terms of patient satisfaction. The aim of this study is to investigate the multi-faceted satisfaction of individuals using assistive devices. Female/male individuals using upper extremity orthosis, lower extremity orthosis, trunk orthosis, lower or upper extremity prosthesis and/or assistive device will be included in the study on a voluntary basis. Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) survey is planned to be used for the evaluation of assistive technology user satisfaction, Orthotics and Prosthetics User's Survey (OPUS) is planned to be used for the evaluation of orthosis prosthesis user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Female/male individuals using upper extremity orthosis, lower extremity orthosis, trunk orthosis, lower or upper extremity prosthesis and/or assistive device
* No cognitive and/or psychological problems
* Individuals without a diagnosis of neurological disease

Exclusion Criteria:

* Diagnosed with a vestibular system disorder
* Diagnosed with a sensorimotor system disorder
* Having an autoimmune disorder
* Individuals with a history of hospitalization for more than three days in the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female individuals using upper extremity orthosis, lower extremity orthosis, trunk orthosis, lower or upper extremity prosthesis and/or assistive devices will be included in the study on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | 5 minute
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) is a survey used to assess the satisfaction of individuals using technological assistive devices. The first version of the survey, developed by Demers et al. in 1996 to assess the satisfaction of using assistive technological devices, consists of 24 items.
Orthotics and Prosthetics Users Survey (OPUS) | 5 minute
  It is preferred to maintain activity development awareness in prosthesis and orthosis applications, to evaluate changes in quality of life, to make quality assessments and to evaluate patients; functional status and satisfaction with prosthesis and orthosis services.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No